CLINICAL TRIAL: NCT01639183
Title: The Effects of Daily Power Toothbrushing on Caregiver Compliance and on Oral and Systemic Inflammation in a Nursing Home Population: A Randomized Controlled Trial
Brief Title: Power Toothbrush Use in Nursing Homes to Eliminate Mouth and Body Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Foundation for Dental Hygiene Research and Education (Other)
Responsible Party: Principal Investigator, Salme E. Lavigne, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H2012:227
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Periodontal Disease
Keywords: oral inflammation; systemic inflammation; compliance; power toothbrushing; nursing home residents
MeSH Terms: conditions — Periodontal Diseases; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotating-oscillating Power Toothbrush (Experimental): Nursing home residents will be randomly assigned to receive power toothbrushing twice daily by their caregivers using a rotating-oscillating power toothbrush.
  Interventions: Device: Rotating-oscillating Power Toothbrush
- Standard Care (Active Comparator): This arm comprises the control group where nursing home residents will receive standard daily oral care as usual.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Rotating-oscillating Power Toothbrush — A power toothbrush will be used twice daily for performing daily oral care on nursing home residents by their caregivers.
  Other Names: Oral-B Professional series 5000 (Proctor & Gamble Co.)
  Arms: Rotating-oscillating Power Toothbrush
Other: Standard Care — Standard daily oral hygiene care by caregivers of nursing home residents whatever that standard care may be.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to investigate whether brushing the teeth of nursing home residents with a power toothbrush as compared with standard care typically provided in nursing homes, will increase caregiver compliance with the provision of daily oral care as well as lower oral and systemic inflammation.

DETAILED DESCRIPTION:
It is well recognized worldwide that residents of nursing homes have poor oral health primarily due to caregiver resistance in the provision of daily oral hygiene care. Fear of being bitten or assaulted by the resident as well as lack of time and discomfort with working in the mouth, are reasons cited for this resistance. It is also now recognized that inflammation in the mouth can raise overall inflammation within the body potentially leading to serious health consequences. Numerous studies involving periodic professional interventions as well as education and training of caregivers in oral care provision have not met with a great deal of success. Caregivers in some studies have indicated preference to power toothbrushes as they are bulkier and longer eliminating the need for insertion of fingers into the mouth and subsequently alleviating fears of being bitten. This study hypothesizes that caregiver utilization of a power toothbrush may increase their compliance with daily oral care provision and could potentially result in elimination of oral and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Nursing Home
* Presence of any natural teeth
* Non-aggressive behavior
* Presence of Periodontal inflammation

Exclusion Criteria:

* Smoking
* Comatose
* On a ventilator
* Aggressive behavior
* Presence of communicable disease
* On antibiotics

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Caregiver Compliance | 6 weeks
  Compliance with power toothbrushing vs standard oral hygiene care will be measured by means of a wall chart filled out by caregivers in the residents rooms.
Systemic Inflammation | 6 weeks
  Systemic inflammation will be measured using a high sensitivity C-reactive protein test (hsCRP. Blood will be drawn at baseline and at 6 weeks to facilitate this test for both intervention and control groups.
Oral Inflammation | 6 weeks
  Oral inflammation will be measured at baseline and 6 weeks by means of 2 tests:
  The Modified Gingival Index (Lobene, 1979) and the Papillary Bleeding Score (Loesche, 1989)

SECONDARY OUTCOMES:
Oral Plaque on Teeth | 6 weeks
  Changes in plaque accumulation on the teeth for both intervention and control groups will be measured using The Turesky Modification (1970) of the Quigley & Hein Plaque Index (1962)

CONTACTS AND LOCATIONS:
Overall Officials: Salme E Lavigne, MS, Principal Investigator — University of Manitoba
Locations (1):
- Deer Lodge Centre, Winnipeg, Manitoba, Canada